CLINICAL TRIAL: NCT04897438
Title: Donor-derived Cell-free DNA for Early Diagnosis of Antibody-mediated Rejection in Kidney Transplant Recipient with Donor-specific Antibodies
Brief Title: Donor-derived Cell-free DNA for Early Diagnosis of Antibody-mediated Rejection
Acronym: cfDNA-DSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Klemens Budde, Senior Physician, Department of Nephrology and Medical Intensive Care, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHA-NTX-001
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Kidney Transplant Rejection; Antibody-mediated Rejection; Kidney Transplant Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Additionally to standard of care, measurements for donor-derived cell-free DNA (dd-cfDNA) are performed at months 0, 1, 3, 6, 9, and 12. If absolute levels of dd-cfDNA are > 50 copies/ml, the patients receive a kidney allograft biopsy. Additionally, kidney allograft biopsies are performed according to standard of care as determined by the treating physicians.
  Interventions: Procedure: Kidney allograft biopsy depending on donor-derived cell-free DNA levels
- Control (No Intervention): Additionally to standard of care, measurements for donor-derived cell-free DNA (dd-cfDNA) are performed at months 0, 1, 3, 6, 9, and 12. These measurements are not used to guide kidney allograft biopsies. Those are performed according to standard of care as determined by the treating physicians.

INTERVENTIONS:
Procedure: Kidney allograft biopsy depending on donor-derived cell-free DNA levels — Kidney allograft biopsy is performed, when absolute levels of donor-derived cell-free DNA are above 50 copies/ml
  Arms: Intervention

SUMMARY:
Patients after kidney transplantation who develop donor-specific antibodies (DSA) are at high risk for antibody-mediated rejection (ABMR). Donor-derived cell-free DNA (dd-cfDNA) levels have been shown to be increased in patients with active or chronic active ABMR. This study aims to evaluate if repeated analysis of dd-cfDNA in patients with DSA and kidney allograft biopsy which is triggered by increased levels of dd-cfDNA can lead to early diagnosis of active or chronic active ABMR among these patients.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years or older
* patients provided written informed consent
* patients after kidney transplantation
* functioning kidney allograft, at least after 180 days after last transplantation
* estimated glomerular filtration rate above 20 ml/min/1.73m^2
* detection of DSA

Exclusion Criteria:

* patients younger than 18 years
* patients unable or did not provide written informed consent
* pregnant or breastfeeding persons
* patients with increased bleeding risk
* patients with multi-organ transplantation
* patients who underwent kidney allograft biopsy after first detection of DSA
* biopsy-proven antibody-mediated rejection
* participation in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Time from study inclusion to diagnosis of antibody-mediated rejection | 12 months after inclusion
  Time from study inclusion date to biopsy-proven diagnosis of active or chronic active antibody-mediated rejection

SECONDARY OUTCOMES:
Sensitivity of absolute dd-cfDNA for detection of ABMR | 12 Months
  Sensitivity of dd-cfDNA > 50 copies/ml to predict the occurence of active or chronic active ABMR in patients with DSA.
Specificity of absolute dd-cfDNA for detection of ABMR | 12 Months
  Specificity of dd-cfDNA > 50 copies/ml to predict the occurence of active or chronic active ABMR in patients with DSA.
Receiver operating characteristics (ROC) analysis of absolute dd-cfDNA for detection of ABMR | 12 Months
  ROC analysis for dd-cfDNA to predict the occurence of active or chronic active ABMR in patients with DSA.
Sensitivity of intraindividual dd-cfDNA changes for detection of ABMR | 12 Months
  Sensitivity of dd-cfDNA increase of > 25% to predict the occurence of active or chronic active ABMR in patients with DSA.
Sensitivity of combined dd-cfDNA criterion for detection of ABMR | 12 Months
  Sensitivity of the combination of "dd-cfDNA increase of > 25%" OR "absolute dd-cfDNA > 50 copies/ml" to predict the occurence of active or chronic active ABMR in patients with DSA.
Clinical Outcome - estimated glomerular filtration rate (eGFR) 12 Months | 12 Months
  Difference between eGFR decline after 12 months between control group and intervention group.
Clinical Outcome - eGFR 24 Months | 24 Months
  Difference between eGFR decline after 24 months between control group and intervention group.
Clinical Outcome - albuminuria 12 Months | 12 Months
  Difference between albuminuria after 12 months between control group and intervention group.
Clinical Outcome - albuminuria 24 Months | 24 Months
  Difference between albuminuria after 24 months between control group and intervention group.
Clinical Outcome - Death-censored Graft Failure 12 Months | 12 Months
  Difference in Death-censored Graft Failure after 12 months between control group and intervention group.
Clinical Outcome - Death-censored Graft Failure 24 Months | 24 Months
  Difference in Death-censored Graft Failure after 24 months between control group and intervention group.
Clinical Outcome - Mortality 12 Months | 12 Months
  Difference in Mortality after 12 months between control group and intervention group.
Clinical Outcome - Mortality 24 Months | 24 Months
  Difference in Mortality after 24 months between control group and intervention group.
Clinical Outcome - Severe Infection 12 Months | 12 Months
  Difference in occurence of severe infections (hospitalization, organ failure, death) during 12 months between control group and intervention group.
Clinical Outcome - Severe Infection 24 Months | 24 Months
  Difference in occurence of severe infections (hospitalization, organ failure, death) during 24 months between control group and intervention group.
Adverse Events of Kidney Transplant Biopsy | 12 Months
  Occurence of Complications from Kidney Transplant Biopsies, including Duration and potential therapy to treat the adverse event.
Rate of ABMR | 12 Months
  Number of biopsy proven active or chronic active ABMR in the cohort.
DSA Levels 0 Months | at inclusion
  Mean fluorescence intensity of immunodominant DSA
DSA Levels 12 Months | 12 months
  Mean fluorescence intensity of immunodominant DSA at 12 months
DSA Levels 24 Months | 24 months
  Mean fluorescence intensity of immunodominant DSA at 24 months
Immunosuppressive Regimen | 24 months
  Report of immunosuppressive medication at the following time points: 0,1,3,6,9,12,24 months, changes of medication, additional therapies such as plasmapheresis, or experimental therapies.
Time from first DSA occurrence to diagnosis of antibody-mediated rejection | 12 months after inclusion
  Time from first DSA occurrence to biopsy-proven diagnosis of active or chronic active antibody-mediated rejection

CONTACTS AND LOCATIONS:
Overall Officials: Klemens Budde, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité-Universitätsmedizin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akifova A, Budde K, Amann K, Buettner-Herold M, Choi M, Oellerich M, Beck J, Bornemann-Kolatzki K, Schutz E, Bachmann F, Halleck F, von Hoerschelmann E, Koch N, Schrezenmeier E, Seelow E, Waiser J, Zukunft B, Eckardt KU, Halbritter J, Kettritz R, Del Moral CL, Lachmann N, Stauch D, Niemann M, Schmidt D, Halloran PF, Osmanodja B. Donor-derived cell-free DNA monitoring for early diagnosis of antibody-mediated rejection after kidney transplantation: a randomized trial. Nephrol Dial Transplant. 2025 Jun 30;40(7):1384-1395. doi: 10.1093/ndt/gfae282. PMID 39673311
- [Derived] Oellerich M, Budde K, Osmanodja B, Bornemann-Kolatzki K, Beck J, Schutz E, Walson PD. Donor-Derived Cell-free DNA for Personalized Immunosuppression in Renal Transplantation. Ther Drug Monit. 2023 Feb 1;45(1):20-25. doi: 10.1097/FTD.0000000000001023. PMID 36127770